CLINICAL TRIAL: NCT06610136
Title: Effects of Acute and Prolonged Caffeine Intake on Neuromuscular Adaptations to Resistance Training in Young Adults
Brief Title: Caffeine and Resistance Training in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEIP2021/6/138
Record Dates: First submitted 2024-09-09; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Caffeine and Resistance Training
MeSH Terms: interventions — Caffeine; Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Caffeine - Males (Experimental)
  Interventions: Dietary Supplement: Caffeine plus Resistance training
- Placebo - Males (Placebo Comparator)
  Interventions: Other: Placebo + Resistance training
- Caffeine - Females (Experimental)
  Interventions: Dietary Supplement: Caffeine plus Resistance training
- Placebo - Females (Placebo Comparator)
  Interventions: Other: Placebo + Resistance training

INTERVENTIONS:
Dietary Supplement: Caffeine plus Resistance training — Acute caffeine intake (3 mg/kg) prior each resistance training session of a 8 weeks training program.
  Arms: Caffeine - Females; Caffeine - Males
Other: Placebo + Resistance training — Acute placebo intake (3 mg/kg of maltodextrin) prior each resistance training session of a 8 weeks training program.
  Arms: Placebo - Females; Placebo - Males

SUMMARY:
Introduction: Several studies have evaluated and confirmed the ergogenic effect of acute caffeine intake on sports performance, specifically on strength and power performance. However, little is known about the prolonged effect of this supplement on neuromuscular adaptations to strength training.

Introduction: Several studies have evaluated and confirmed the ergogenic effect of acute caffeine intake on sports performance, specifically on strength and power performance. However, little is known about the prolonged effects of this supplement on neuromuscular adaptations to strength training.

Objectives: The present study aims to analyze the effects of acute and chronic caffeine intake on neuromuscular adaptations to strength training, according to sex (men vs. women) and type of exercise (bench press vs. squat), as well as on fatigue resistance during repeated sprints, fatigue perception, mood state, reaction time, diet, and potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 18 and ≤ 35 years.
* Body mass index (BMI) < 25 kg/m².
* Physically active subjects (>150 min/week of moderate exercise).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from performing physical exercise.
* Participants capable of performing the tests.

Exclusion Criteria:

* History of neuromuscular, cardiac, or diseases that could affect liver or muscle metabolism.
* Use of drugs or other stimulants that interfere with caffeine intake and intestinal absorption during the tests and study.
* Body mass index (BMI) > 25 kg/m².
* Having undergone prolonged periods of forced physical inactivity during the 6 months prior to the study.
* Performing strenuous exercise within 48 hours prior to the tests.
* Failing to replicate the same food intake on the two experimental days.
* Consuming caffeine after 6 PM on the day prior to training or testing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Mean velocity at different %1RM | Through study completion, an average of 12 weeks
  Measuring bar mean velocity desplacement during bench press and back squat exercises.
Peak velocity at different %1RM | Through study completion, an average of 12 weeks
  Measuring bar peak velocity and time to reach peak velocity of bar desplacement during bench press and back squat exercises.
Mean power output at different %1RM | Through study completion, an average of 12 weeks
  Measuring during bench press and back squat exercises.
Peak power output and time to reach peak power output at different %1RM | Through study completion, an average of 12 weeks
  Measuring during bench press and back squat exercises.
Number of repetitions performed at 65%1RM until task failure | Through study completion, an average of 12 weeks
  In bench press and back squat exercises
Bar velocity deplacement performed in 1 set at 65%1RM until task failure | Through study completion, an average of 12 weeks
  In bench press and back squat exercises
Power output generated in 1 set at 65%1RM until task failure | Through study completion, an average of 12 weeks
  In bench press and back squat exercise

SECONDARY OUTCOMES:
Resting Metabolic Rate (RMR) | Through study completion, an average of 12 weeks
  Kcal at rest using a metabolic chart.
Maximal Fat Oxidation Rate (MFO) | Through study completion, an average of 12 weeks
  g/min using a metabolic chart.
Fat mass | Through study completion, an average of 12 weeks
  Using electrical bioimpedance (kg and % of body mass)
Fat-free mass | Through study completion, an average of 12 weeks
  Using electrical bioimpedance (kg and % of body mass)
Physical activity (METs-min/wk) | Through study completion, an average of 12 weeks
  Using IPAQ
Dietary (g/kg of macronutrients) | Through study completion, an average of 12 weeks
  Using a 24-total recall
Mood state | Through study completion, an average of 12 weeks
  Mood. Participants graded a set of 29 items related to the mood on a Likert scale from 0 (not at all) to 4 (extremely) in reply to the question;How do you feel at this moment?; to assess six scales: tension, depression, anger, vigor, fatigue and confusion.
Adverse effects | Through study completion, an average of 12 weeks
  Adverse effects. perception of power, endurance, energy and exertion, as well as heart, muscular and gastrointestinal discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes